CLINICAL TRIAL: NCT01821170
Title: Cognitive Remediation in ADHD Children : Comparison Between Three Therapeutic Strategies : Cognitive Remediation With a Virtual Classroom Software and Methylphenidate and Supportive Psychotherapy
Acronym: RECOGNITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Fondation Caisse d'Epargne (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2012/16
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: ADHD
Keywords: ADHD; children; cognitive remediation; virtual reality
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive remediation (Experimental)
  Interventions: Device: cognitive remediation; Other: neuropsychological tests
- Supportive psychotherapy (Active Comparator)
  Interventions: Behavioral: supportive psychotherapy; Other: neuropsychological tests
- Methylphenidate (Active Comparator)
  Interventions: Drug: Methylphenidate; Other: neuropsychological tests

INTERVENTIONS:
Drug: Methylphenidate — Patient will take treatment during two months
  Arms: Methylphenidate
Device: cognitive remediation — Patient will have 12 sessions during 6 to 8 weeks
  Arms: Cognitive remediation
Behavioral: supportive psychotherapy — Patients will have 12 sessions during 6 to 8 weeks
  Arms: Supportive psychotherapy
Other: neuropsychological tests — neuropsychological tests will assess attentional and executive performance

SUMMARY:
The Attention Deficit Disorder with or without Hyperactivity (ADHD) is one of the most frequently found disorder in children. It is characterized by a triad of symptoms involving attention deficit, hyperactivity and impulsivity and having an impact on the functioning of the subject especially in terms of learning.

Currently, main interventions to treat ADHD in children are stimulant medication or supportive psychotherapy. Data from recent studies highlight the use of stimulant drugs (amphetamine derivatives such as methylphenidate) to treat the core symptoms of ADHD children. These drugs are generally effective but their nature (psychostimulants) and adverse effects they cause (appetite suppression, sleep disturbances, headaches, motor tics, abdominal pain, irritability, nausea and fatigue) encourage the development of new therapeutic approaches. The use of supportive psychotherapy alone would have limited effect on symptoms of children with ADHD. Our aim is to test the use a cognitive remediation program using a virtual classroom in children suffering from ADHD.

DETAILED DESCRIPTION:
Virtual reality offers the possibility to develop environments approaching situations of daily life that can be used to target evaluation but also for therapeutic purposes. As the school classroom is a daily life situation for children, Rizzo team has developed a virtual classroom software (Rizzo et al., 2006). This virtual classroom is a tool for the diagnosis of ADHD based on the exploration of attention deficit (distractibility, sustained attention ...), impulsivity and hyperactivity. On the other hand, the playfulness of the application helps the child to "forget" quickly that he is placed in a test situation.

In the virtual classroom, the requested task is a letter detection task. The subject had to click on the mouse only when he sees the letter "K" preceded by the letter "A" appearing. The child had to perform this task, while the disruptive elements are distracting. These may be auditory (the bell ringing), visual (a paper airplane flying in the class) or visual and auditory distractors (the sound of the teacher who is moving).

Cognitive remediation using virtual reality is an innovative approach in the care of children. We want to examine whether a cognitive remediation program based on the virtual classroom software can be a therapeutic tool for children suffering from ADHD.

In our study, cognitive remediation will be accomplished through cognitive intervention such as a "training" of attentional and executive functions (such as planning, working memory, selective attention, ...). The cognitive remediation sessions will include the execution of the virtual classroom protocol, a stage of metacognition and again the virtual classroom assessment. Our remediation program will include 12 sessions (twice a week for 6 to 8 consecutive weeks), lasting 30 minutes each. The effects of cognitive remediation will be compared to the effects of two other major interventions usually proposed: drug treatment with methylphenidate and supportive psychotherapy. 60 ADHD children aged 7 to 11 years will participate in our study, 20 in each treatment group (drug treatment vs. cognitive remediation vs. supportive psychotherapy).

We expect that cognitive remediation and drug treatment improve attentional abilities of children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 7 to 11 years,
* Responding to current diagnostic criteria for ADHD according to DSM IV-TR (Diagnostic and Statistical Manual of Mental Disorders),
* Presenting a total score on the ADHD-RS (ADHD Rating Scale)> 28 (before treatment),
* Schooled in conventional class,
* Presenting a WISC (Wechsler Intelligence Scale for Children) IV total score> 80 (done before or in follow-up),
* Registered to social security,
* Legal represent has given informed consent to participate in the study.

Exclusion Criteria:

* Uncorrected perceptual disorder,
* Patient treated by psychostimulant,
* Patient under supportive psychotherapy,
* Patient treated by methylphenidate,
* Subjects with a pervasive developmental disorder, psychotic disorder, characterized major depressive disorder,
* Subjects who participated in research in the last 3 months,
* Subjects suffering from: glaucoma, hyperthyroidism, thyrotoxicosis, heart diseases (high blood pressure, congestive heart failure, etc…), cerebrovascular disorders,
* Subjects with no deficit in the virtual classroom: having a total number of hit superior to 80 and a number of commissions inferior to 21.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2016-04-27 (Actual)

PRIMARY OUTCOMES:
Score at ADHD Rating Scale before and after treatment | At the end of study (week 8 after inclusion)

SECONDARY OUTCOMES:
Performance of participants in neuropsychological tests assessing executive and attentional abilities before and after treatment | At the end of study (week 8 after inclusion)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie BIOULAC, MD, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Charles Perrens, Bordeaux